CLINICAL TRIAL: NCT01953107
Title: A Randomized Controlled Trial of Pre-Operative Treatment With Ferrous Fumarate 300 mg Once Daily Versus Placebo in Newly Diagnoses Gynecologic Oncology Patients Who Are Primary Surgical Candidates.
Brief Title: Oral Iron vs. Placebo in Newly Diagnosed Gynecologic Oncology Patients Who Are Surgical Candidates.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Danielle Vicus, Surgical Oncologist - Gynecologic Oncology, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GYNEOCC2
Record Dates: First submitted 2013-08-26; First posted 2013-09-30 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Ovarian Cancer; Cervical Cancer; Uterine Cancer; Anemia
Keywords: Anemia; Ovarian cancer; Uterine cancer; Cervical cancer; Oral iron
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Cervical Neoplasms; Uterine Neoplasms; Anemia | interventions — ferrous fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferrous Fumarate 300 mg + Vitamin C (Experimental): 300 mg once a day of Oral Ferrous Fumarate
  Interventions: Other: Oral Ferrous Fumarate
- Placebo + Vitamin C (Placebo Comparator): 300 mg of Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Oral Ferrous Fumarate
  Arms: Ferrous Fumarate 300 mg + Vitamin C
Other: Placebo
  Arms: Placebo + Vitamin C

SUMMARY:
The prevalence of anemia in gynecologic oncology new patients has been seen in previous studies to be as high as 35-59%. this population includes women with several types of gynecologic malignancies. Therefore, it is assumed that the origin of the anemia can be due to anemia of chronic disease and iron deficiency anemia. No previous studies have looked at the efficacy of oral iron supplementation with concurrent Vitamin C in women with newly diagnosed gynecologic malignancies.

Hypothesis: In newly diagnosed gynecologic oncology patients who are surgical candidates does treatment with 3-6 weeks of oral ferrous fumarate 300 mg once a day improve the mean change in hemoglobin levels, from baseline to pre-operative, in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Scheduled for primary operative procedure within 3-6 weeks of initial consult clinic visit with endometrial cancer, uterine sarcoma, cervical cancer, ovarian/fallopian tube cancer or patients with pelvic mass and a high suspicion of a gynecologic malignancy.

Exclusion Criteria:

* Patient with known allergy to ferrous fumarate.
* Patient's on IV Iron or erythropoietin treatment at the time of recruitment
* Patient's who are not primary surgical candidates.
* Patient's with a known hemoglobinopathy or a hypoproliferative hematologic disorder
* Patient who have significant active vaginal bleeding
* Patient who have a hemoglobin < 80 g/L will be removed from randomization and referred to blood conservation at Sunnybrook Health SCiences Centre.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-01 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Mean Difference in Hemoglobin | Pre-surgery (4-6 weeks)
  The mean difference in the change of hemoglobin levels from baseline to the day of surgery between participants treated with oral iron versus. placebo.

SECONDARY OUTCOMES:
Quality of life | Baseline to Pre-surgery (4-6 weeks)
  The difference in quality of life (FACT-An) between patients treated with ferrous fumarate 300 mg. daily to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Vicus, MD, Principal Investigator — Odette Cancer Centre
Locations (1):
- Odette Cancer Centre, Toronto, Ontario, Canada